CLINICAL TRIAL: NCT03399552
Title: An Efficacy and Safety Study of Avelumab Plus SBRT in Malignant Mesothelioma (MPM)
Brief Title: Stereotactic Body Radiation Therapy and Avelumab Immunotherapy for Treatment of Malignant Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-358
Record Dates: First submitted 2018-01-09; First posted 2018-01-16 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-01

CONDITIONS: Malignant Mesothelioma (MPM)
Keywords: Stereotactic Body Radiation Therapy; Avelumab Immunotherapy; 17-358
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — avelumab; Radiosurgery

STUDY DESIGN:
Intervention Model Description: This is a single-arm, two-stage study that will be conducted at Memorial Sloan Kettering Cancer Center Main Campus and regional sites.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): The treatment will consist of one dose of avelumab every other week as well as a short course of SBRT after the first two doses of avelumab.
  Interventions: Drug: Avelumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Avelumab — 10mg/kg delivered by IV infusion
Radiation: Stereotactic Body Radiation Therapy — short course of SBRT after the first two doses of avelumab

SUMMARY:
The purpose of this study is to find out whether the combination of avelumab and SBRT is safe and what effect avelumab has on mesothelioma when given in combination with SBRT. In addition, a goal of this protocol is to study the effect of radiation therapy on the immune system. It is thought that radiation treatment may create a form of 'vaccine' against cancer inside the body and immunotherapy may improve this effect. The combination of radiation treatment and immunotherapy may be more effective against cancer than either radiation or immunotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to provide written informed consent for the trial.
* Patient age ≥ 18 at time of consent.
* Histologically or cytologically confirmed malignant pleural or peritoneal mesothelioma (MPM).
* No plans for surgical resection.
* At least one prior line of systemic therapy. Note: Patients on prior immunotherapy are eligible.
* At least one targetable lesion appropriate for palliative SBRT and one non-target lesion
* Karnofsky Performance Score (KPS) ≥ 70%
* If of childbearing potential, must be willing to use highly effective mode of contraception for at least one month prior, during, and for 2 months after the end of active therapy
* Adequate organ function, defined as:

  * Absolute Neutrophil Count ≥ 1.5K/mcL.
  * Platelet count ≥ 100K/mcL.
  * Adequate renal function as defined by an estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula or serum creatinine ≤ 1.5 x ULN
  * Hemoglobin > 9g/dL (prior transfusion permitted)
  * Total bilirubin level ≤ 1.5 × the upper limit of normal (ULN) range
  * AST and ALT levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver).
* If the patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

Exclusion Criteria:

* Currently participating and receiving another study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Prior radiation therapy precluding SBRT
* Continuous oxygen use
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* Patient who rapidly progressed on prior immunotherapy, as determined by the treating physician, are not eligible.
* Prior Therapies:

  1. Treatment with a monoclonal antibody within 4 weeks prior to study Day 1 or has not recovered (i.e., ≥ Grade 1 at baseline) from adverse events due to agents administered
  2. Prior chemotherapy, targeted small molecule therapy, within 4 weeks prior to study Day 1 or has not recovered (i.e., ≥ Grade 1 at baseline) from adverse events due to a previously administered agent (excluding Grade 2 neuropathy).
  3. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) within 4 weeks prior to study Day 1 or has not recovered (i.e., >/= Grade 1 at baseline) from adverse events
* Comorbidities or Prior Conditions:

  1. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  2. Prior organ transplantation including allogenic stem-cell transplantation.
  3. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
  4. Known history of active TB (Tuberculosis).
  5. Known history of HIV or known acquired immunodeficiency syndrome.
  6. Active Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection at screening or positive serologies indicating prior infection.
  7. Active infection requiring systemic therapy.
  8. Evidence of interstitial lung disease or active, non-infectious pneumonitis.
  9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Pregnant women or women who are breastfeeding or of childbearing potential and not using a highly effective method of birth control for at least one month prior to enrollment. If the risk of contraception exists, male and female subjects must use highly effective contraception throughout the study and for at least 60 days after last avelumab treatment.

  a. Highly effective contraception includes either 2 barrier methods (diaphragm, condom by the partner, copper intrauterine device, sponge, or spermicide), or 1 barrier method and 1 hormonal method (any oral, subcutaneous, intrauterine, or intramuscular registered and marketed contraceptive agent that contains an estrogen and/or a progesterone agent).
* Vaccination within 4 weeks prior to the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.
* Concomitant use of the following medications

  1. Any investigational anticancer therapy.
  2. Any concurrent chemotherapy, immunotherapy, or biologic therapy. Concurrent use of hormones for non-cancer-related conditions (e.g., insulin for diabetes and hormone replacement therapy) is acceptable.
  3. Immunosuppressive medications including, but not limited to systemic corticosteroids (>10 mg/day prednisone or equivalent), methotrexate, azathioprine, and tumor necrosis factor alpha (TNF-α) blockers. Use of immunosuppressive medications for the management of investigational product-related AEs, in subjects with contrast allergies is acceptable. In addition, use of inhaled and intranasal corticosteroids is permitted.
* Known contraindications to radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Rimner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Avelumab: The treatment will consist of avelumab as well as a short course of Stereotactic Body Radiation Therapy
Period: Overall Study
Arm/Group | Avelumab
Started | 15
Completed | 13
Not Completed | 2
Not completed — No evidence of disease | 1
Not completed — Unevaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 71 [51 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: defined by modified RECIST 1.1 for mesothelioma
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 15
Participants
  Clinical Progression | 2
  Stable Disease | 8
  Partial Response | 1
  Non-evaluable | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 14/15
Serious Adverse Events (participants affected / at risk) | 14/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=15)
Death due to disease progression (General disorders) | 2
Death NOS (General disorders) | 12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab (N=15)
Infusion-related allergic reactions (Injury, poisoning and procedural complications) | 6
Anorexia (Metabolism and nutrition disorders) | 6
Fatigue (General disorders) | 6
Thyroid disorders (Endocrine disorders) | 5
Diarrhea (Gastrointestinal disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT03399552/Prot_SAP_000.pdf